CLINICAL TRIAL: NCT00732784
Title: Effect of Calcium Supplements on Imatinib Mesylate (Gleevec®) Pharmacokinetics in Healthy Volunteers (CSTI571BUS 280) (UPCI 08-072)
Brief Title: Effect of Calcium on Gleevec Pharmacokinetics (PK) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jan Beumer (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jan Beumer, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 08-072; CSTI571BUS 280; UPCI 08-072
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Healthy volunteers; No condition; Pharmacokinetics study
MeSH Terms: interventions — Imatinib Mesylate; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): On an 18-day schedule, calcium supplement (Tums Ultra 1000®) once daily on day 15; and Gleevec® once daily on days 1 and 15 (i.e., Gleevec® alone on day 1, and combination of Gleevec® and calcium supplement on day 15).
  Interventions: Drug: Imatinib mesylate; Dietary Supplement: calcium carbonate
- 2 (Other): On an 18-day schedule, calcium supplement (Tums Ultra 1000®) once daily on day 1; and Gleevec® once daily on days 1 and 15 (i.e., combination of Gleevec® and calcium supplement on day 1, Gleevec® alone on day 15).
  Interventions: Drug: Imatinib mesylate; Dietary Supplement: calcium carbonate

INTERVENTIONS:
Drug: Imatinib mesylate — Dosage form: tablets Dosage: 400 mg Frequency & duration: On an 18-day schedule, one dose administered once on day 1 and once on day 15 (2 doses total)
  Other Names: Gleevec®; STI571
Dietary Supplement: calcium carbonate — Dosage form: tablets Dosage: 4000 mg (4 x 1000 mg tablet) Frequency: On an 18-day schedule, once daily day 15 (for Arm 1); or once daily day 1 (for Arm 2)
  Other Names: Tums Ultra 1000®

SUMMARY:
This research study is being conducted through the University of Pittsburgh Cancer Institute (UPCI). It will evaluate the concentrations of Gleevec®, an oral drug used to treat some types of cancer, in the blood of healthy volunteers when taken with and without Tums Ultra®, a calcium product often used in the treatment of upset stomach and as a calcium supplement.

DETAILED DESCRIPTION:
This is an open-label, single-institution, randomized cross-over, fixed-schedule investigation of the effects of calcium carbonate on the pharmacokinetics (PK) of Gleevec® in healthy volunteers. Healthy volunteers will be recruited to participate in this study such that twelve subjects (6 men / 6 women) will complete the study at UPCI. Subjects will be compensated for participation.

Half of the subjects will receive Gleevec® alone on Day 1 and Gleevec® and calcium carbonate on Day 15, and the other half will receive Gleevec® and calcium carbonate on Day 1 and Gleevec® alone on Day 15, determined by randomization of subjects receiving either the combination or Gleevec® alone during the first visit. Doses will be 400 mg Gleevec® and 4000 mg calcium carbonate (4 x Tums Ultra 1000® chewable tablets, equivalent to 4000 mg calcium carbonate or 1600 mg calcium.

Multiple PK blood samples will be taken from Days 1-4 and Days 15-18. Gleevec® PK will be assessed after oral administration of 400 mg Gleevec® alone, and after oral administration of 400 mg Gleevec® with concomitant administration of 4000 mg calcium carbonate. Two 10-hour outpatient dosing visits and six brief outpatient visits are required to accommodate all study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women 18 years of age or older. Healthy subjects are defined as individuals who are free from clinically significant illness or disease (such as coronary arterial disease, chronic heart failure, bleeding disorder, hypertension, chronic renal failure etc.) as determined by their medical history, physical examination, and laboratory studies. For the purposes of this protocol, "clinically significant" is defined as any history or indication of illness or disease, such as those listed above.
* Body Mass Index (BMI) < 31 kg/m2 (weight/height2).
* Female patients of childbearing potential must have negative pregnancy test within 14 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 7 days following discontinuation of study drug.
* Written, voluntary informed consent.

Exclusion Criteria:

* Abnormal marrow function as defined by leucocyte, neutrophil, or platelet counts outside of normal limits.
* Any evidence of renal dysfunction (proteinuria; serum creatinine > upper limit of normal; or if serum creatinine > upper limit of normal, a calculated creatinine clearance < 60 mL/min/1.73 m2).
* Impaired hepatic function (liver enzymes greater than the upper limit of normal or bilirubin outside the normal range).
* Taking any medications (including over the counter products), herbal products, mineral supplements or vitamins (other than a daily multivitamin preparation), other than contraceptives (for women), within 2 weeks of start of the study. All forms of contraceptive medication are permissible for this study and would not result in a female's exclusion from participation. Patients who take medications on a chronic basis, such as antihypertensive medications or thyroid replacement therapy, etc. are not eligible for the study.
* Subjects has received any other investigational agents within 28 days of first day of study drug dosing.
* Female subjects who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To define the effect of administration of a calcium salt (calcium carbonate) on the PK (in particular the area under the imatinib plasma concentration versus time curve) of imatinib (Gleevec®) in healthy volunteers. | PK blood samples are drawn from each subject at time 0 (before each dose of Gleevec®), and at 0.5, 1, 2, 3, 4, 5, 6, 8, 24, 48, and 72 hrs after adminstration of Gleevec®.

CONTACTS AND LOCATIONS:
Overall Officials: Jan H. Beumer, PharmD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute / Clinical and Translational Research Center (Hillman Cancer Center location), Pittsburgh, Pennsylvania, United States